CLINICAL TRIAL: NCT02279394
Title: E- PRISM: Precision Intervention Smoldering Myeloma: Phase II Trial of Combination of Elotuzumab, Lenalidomide and Dexamethasone in High-Risk Smoldering Multiple Myeloma
Brief Title: E-PRISM: Phase II Trial of Elotuzumab Lenalidomide and Dexamethasone in High-Risk Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Celgene (Industry); Blood Cancer Research Partnership (Other); Multiple Myeloma Research Consortium (Network); The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-338
Record Dates: First submitted 2014-09-26; First posted 2014-10-31 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Smoldering Myeloma; Smoldering Multiple Myeloma
Keywords: Smoldering myeloma; Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elo / Len / Dex (Experimental): •Drug: Elotuzumab 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Other Name: HuLuc63
  •Drug: Lenalidomide 25 mg Oral; Days 1-21 days Cycles 1-24
  Other Name: REVLIMID
  •Drug: Dexamethasone 40 mg Oral; Days 1, 8, 15, 22 Cycles 1-2 40 mg Oral; Days 1, 8, 15 Cycles 3-8
  Other Name: Decadron
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide; Drug: Dexamethasone
- Elo / Len (Experimental): •Drug: Elotuzumab 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Other Name: HuLuc63
  •Drug: Lenalidomide 25 mg Oral; Days 1-21 days Cycles 1-24
  Other Name: REVLIMID
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Elotuzumab — 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Other Names: HuLuc63
Drug: Lenalidomide — 25 mg Oral; Days 1-21 days Cycles 1-24
  Other Names: REVLIMID
Drug: Dexamethasone — 40 mg Oral; Days 1, 8, 15, 22 Cycles 1-2 40 mg Oral; Days 1, 8, 15 Cycles 3-8
  Other Names: Decadron
  Arms: Elo / Len / Dex

SUMMARY:
This research study is aimed to determine the proportion of high risk smoldering multiple myeloma patients who are progression free at 2 years after receiving elotuzumab, lenalidomide and dexamethasone combination therapy.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial, which tests the effectiveness of the investigational drugs elotuzumab, lenalidomide and dexamethasone in smoldering multiple myeloma. Recent research studies have shown that early treatment of smoldering multiple myeloma may delay or prevent the progression to active multiple myeloma. The purpose of this research study is to learn whether the combination of elotuzumab, lenalidomide and dexamethasone works in treating smoldering multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Must have smoldering myeloma with high risk markers based on the Mayo OR the Spanish criteria as described below
* >10% plasma cells in the bone marrow and any one or more of the following:

  * Serum M protein of 3 g/dL or greater
  * IgA SMM
  * Immunoparesis with reduction of two uninvolved immunoglobulin isotypes
  * Serum involved/uninvolved free light chain ratio ≥8 (but less than 100)
  * Progressive increase in M protein level (Evolving type of SMM)†
  * Bone marrow clonal plasma cells 50-60%
  * Abnormal plasma cell immunophenotype (≥95% of bone marrow plasma cells are clonal) and reduction of one or more uninvolved immunoglobulin isotypes
  * t (4;14) or del 17p or 1q gain
  * Increased circulating plasma cells
  * MRI with diffuse abnormalities or 1 focal lesion
  * PET-CT with focal lesion with increased uptake without underlying osteolytic bone destruction † Increase in serum monoclonal protein by ≥25% on two successive evaluations within a 6 month period
* No evidence of CRAB (see below for details) criteria or new criteria of active multiple myeloma which including the following:

  * Increased calcium levels (corrected serum calcium >0.25 mmol/dL above the upper limit of normal or >.275 mmol/dL)
  * Renal insufficiency (attributable to myeloma)
  * Anemia (Hb 2g/dL below the lower limit of normal or <10g/dL)
  * Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
  * No evidence of the following new criteria for active MM including the following: Bone marrow plasma cells ≥ 60%, Serum involved/uninvolved FLC ratio ≥100, and MRI with more than one focal lesion

    * Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible
* ECOG Performance Status (PS) 0, 1, or 2 (Appendix A)
* The following laboratory values obtained ≤ 14 days prior to registration:

  * ANC ≥1000/µL
  * PLT ≥ 50,000/µL
  * Total bilirubin ≤ 2.0 mg/dL (If total is elevated check direct and if normal patient is eligible.)
  * AST ≤ 3 x institutional upper limit of normal (ULN)
  * ALT ≤ 3 x institutional upper limit of normal (ULN)
  * Estimated creatinine clearance ≥ 60mL/min or a creatinine ≤ 2.2 mg/dL
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Females of childbearing potential* must have a negative serum or urine pregnancy test
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy
* Ability to understand and the willingness to sign a written informed consent.
* Exclusion Criteria:
* Symptomatic Multiple Myeloma or any evidence of CRAB criteria including the new criteria for overt myeloma. Any prior therapy for active Myeloma should also be excluded. Prior therapy for smoldering myeloma is not an exclusion criteria. Bisphosphonates are not excluded
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational. Prior therapy with bisphosphonate is allowed. Prior radiation therapy to a solitary plasmacytoma is allowed. Prior clinical trials for smoldering MM or MGUS are allowed as long as the last therapy was at least 2 months prior and there was no improvement in M spike
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Uncontrolled intercurrent illness
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to elotuzumab or lenalidomide
* Known seropositive for or active viral infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus. Patients who are seropositive because of hepatitis B virus vaccine are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - St Francis Hospital and Medical Center, Hartford, Connecticut
  - University of Chicago, Chicago, Illinois
  - Eastern Maine Medical Center, Brewer, Maine
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Levine Cancer Institute, Charlotte, North Carolina

REFERENCES:
- [Derived] Kazandjian D, Diamond B, Papadimitriou M, Hill E, Sklavenitis-Pistofidis R, Ziccheddu B, Blaney P, Chojnacka M, Durante M, Maclachlan K, Young R, Usmani S, Davies F, Getz G, Ghobrial I, Korde N, Morgan G, Maura F, Landgren O. Genomic Profiling to Contextualize the Results of Intervention for Smoldering Multiple Myeloma. Clin Cancer Res. 2024 Oct 1;30(19):4482-4490. doi: 10.1158/1078-0432.CCR-24-0210. PMID 38652812

RESULTS

PARTICIPANT FLOW:
Groups:
- Elo / Len / Dex: •Drug: Elotuzumab 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Other Name: HuLuc63
  •Drug: Lenalidomide 25 mg Oral; Days 1-21 days Cycles 1-24
  Other Name: REVLIMID
  •Drug: Dexamethasone 40 mg Oral; Days 1, 8, 15, 22 Cycles 1-2 40 mg Oral; Days 1, 8, 15 Cycles 3-8
  Other Name: Decadron
  Elotuzumab: 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Lenalidomide: 25 mg Oral; Days 1-21 days Cycles 1-24
  Dexamethasone: 40 mg Oral; Days 1, 8, 15, 22 Cycles 1-2 40 mg Oral; Days 1, 8, 15 Cycles 3-8
- Elo / Len: •Drug: Elotuzumab 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Other Name: HuLuc63
  •Drug: Lenalidomide 25 mg Oral; Days 1-21 days Cycles 1-24
  Other Name: REVLIMID
  Elotuzumab: 10 mg/kg IV; Days 1, 8,15, 22 Cycles 1-2 10 mg/kg IV; Days 1 & 15 Cycles 3-8
  Lenalidomide: 25 mg Oral; Days 1-21 days Cycles 1-24
Period: Overall Study
Arm/Group | Elo / Len / Dex | Elo / Len
Started | 40 | 11
Completed | 40 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elo / Len / Dex | Elo / Len | Total
Number analyzed (Participants) | 40 | 11 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 8 | 31
  >=65 years | 17 | 3 | 20
Age, Continuous [Median (Full Range); unit: years] | 62 [29 to 79] | 62 [44 to 75] | 62 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 6 | 32
  Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 37 | 11 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 31 | 11 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 11 | 51
ECOG Performance Status [Count of Participants; unit: Participants] — 0 = Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  1= Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  2 = In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    00 - Fully Active | 27 | 7 | 34
    01 - Restricted | 12 | 4 | 16
    02 - Ambulatory | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Are Progression Free at 2 Years
Description: Percent of patients who are alive and without documented progression after at least 2-years of follow-up. All patients who receive study treatment are assessed including those who have died or lost to follow-up prior to 2-years. Progression was defined as an increase in SPEP [25% and an absolute increase of 0.5g/d] or UPEP [25% and an absolute increase of 200mg/24hours] on 2 successive evaluations as determined by the IMWG response criteria or documented progression by the FreeLite progressive disease criteria in the absence of serum or urine involvement.
Time Frame: 2 Years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Elo / Len / Dex | Elo / Len
Number analyzed (Participants) | 40 | 11
percentage of participants | 45.0 [31.5 to 59.1] | 36.4 [13.6 to 65.0]

2. Secondary Outcome: Objective Response Percent
Description: Percent of patients with objective response defined as partial response or better based on the International Myeloma Working Group Response (IMWG) criteria
Time Frame: 2 Years from start of treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Elo / Len / Dex | Elo / Len
Number analyzed (Participants) | 40 | 11
percentage of participants | 82.5 [69.6 to 91.5] | 72.7 [43.6 to 92.1]

3. Secondary Outcome: Time to Progression
Description: Time from initiation of therapy to progression defined by the IMWG criteria.
Time Frame: From start of treatment up to +/- 60 months
Measure: Median (Full Range); unit: months
Arm/Group | Elo / Len / Dex | Elo / Len
Number analyzed (Participants) | 40 | 11
months | 56.1 [9.3 to 61.4] | 56.2 [27.9 to 62.5]

4. Secondary Outcome: Overall Survival
Description: Time from initiation of therapy to death
Time Frame: From start of treatment up to +/- 60 months
Measure: Median (Full Range); unit: months
Arm/Group | Elo / Len / Dex | Elo / Len
Number analyzed (Participants) | 40 | 11
months | 50.5 [11.3 to 61.4] | 60.2 [39.1 to 66.0]

ADVERSE EVENTS:
Time Frame: Adverse Events assessed/monitored from the day of consent up to the end of treatment for an average of 26 months All-Cause Mortality as well as Serious Adverse Events were collected up to +/- 60 months. These duration may vary individually based on possible dose delays as well as follow up study visit delays or some participants possibly coming off study early.
Arm/Group | Elo / Len / Dex | Elo / Len
All-Cause Mortality (participants affected / at risk) | 2/40 | 0/11
Serious Adverse Events (participants affected / at risk) | 8/40 | 1/11
Other Adverse Events (participants affected / at risk) | 40/40 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elo / Len / Dex (N=40) | Elo / Len (N=11)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Myocardial infarction (General disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hypophosphatemia (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elo / Len / Dex (N=40) | Elo / Len (N=11)
Fatigue (General disorders) | 36 (72) | 11 (47)
Diarrhea (Gastrointestinal disorders) | 32 (70) | 6 (24)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (82) | 9 (43)
White blood cell decreased (Investigations) | 22 (97) | 5 (11)
Insomnia (Psychiatric disorders) | 21 (28) | 5 (7)
Nausea (Gastrointestinal disorders) | 20 (29) | 5 (17)
Anemia (Blood and lymphatic system disorders) | 17 (48) | 6 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 18 (78) | 8 (26)
Upper respiratory infection (Infections and infestations) | 18 (33) | 5 (11)
Constipation (Gastrointestinal disorders) | 16 (29) | 6 (16)
Neutrophil count decreased (Investigations) | 19 (131) | 4 (28)
Platelet count decreased (Investigations) | 17 (71) | 3 (16)
Hypokalemia (Metabolism and nutrition disorders) | 10 (25) | 7 (20)
Hypomagnesemia (Metabolism and nutrition disorders) | 13 (28) | 3 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (31) | 5 (23)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (17) | 3 (6)
Lymphocyte count decreased (Investigations) | 12 (76) | 2 (22)
Hyponatremia (Metabolism and nutrition disorders) | 8 (22) | 4 (14)
Aspartate aminotransferase increased (Investigations) | 8 (14) | 3 (5)
Anxiety (Psychiatric disorders) | 7 (7) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (19) | 1 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 1 (1)
Edema limbs (General disorders) | 6 (9) | 3 (3)
Headache (Nervous system disorders) | 7 (10) | 2 (8)
Hypertension (Vascular disorders) | 8 (17) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (14) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (9) | 3 (5)
Alanine aminotransferase increased (Investigations) | 6 (10) | 2 (2)
Dizziness (Nervous system disorders) | 6 (11) | 2 (4)
Dysgeusia (Nervous system disorders) | 7 (7) | 1 (1)
Fever (General disorders) | 7 (11) | 1 (2)
Lung infection (Infections and infestations) | 8 (9) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (3) | 4 (5)
Depression (Psychiatric disorders) | 5 (5) | 1 (2)
Infections and infestations - Other (Infections and infestations) | 5 (6) | 1 (2)
Infusion related reaction (General disorders) | 4 (4) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 3 (5)
Sinusitis (Infections and infestations) | 5 (7) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Agitation (Psychiatric disorders) | 4 (4) | 1 (2)
Alkaline phosphatase increased (Investigations) | 3 (6) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Flu like symptoms (General disorders) | 5 (6) | 0 (0)
Hypotension (Vascular disorders) | 5 (7) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Skin/subcutaneous tissue disorders; Other (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Thromboembolic event (Vascular disorders) | 4 (4) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (7)
Blurred vision (Eye disorders) | 4 (5) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Weight gain (Investigations) | 3 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Bloating (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 2 (3)
Pain (General disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02279394/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT02279394/ICF_001.pdf